CLINICAL TRIAL: NCT01416714
Title: Tissue Procurement for Gastric Cancer, Gastrointestinal Stromal Tumors (GIST), Esophageal Cancer, Pancreas Cancer, Hepatocellular Cancer, Biliary Cancer, Neuroendocrine, Peritoneal Mesothelioma, Anal Cancer and Colorectal Cancer in Patients Undergoing Surgery or Biopsy
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 16294A
Record Dates: First submitted 2010-08-20; First posted 2011-08-15 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancers
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, tissue, DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (10):
- Gastric Cancer
- Gastrointestinal Stromal Tumors (GIST)
- Esophageal Cancer
- Pancreas Cancer
- Hepatocellular Cancer
- Biliary Cancer
- Neuroendocrine Cancer
- Peritoneal Mesothelioma
- Anal Cancer
- Colorectal Cancer

SUMMARY:
The purpose of this study is to collect and store normal and malignant tissue from patients with gastric cancer, GIST, esophageal cancer, pancreas cancer, hepatocellular cancer, biliary cancer, neuroendocrine, peritoneal mesothelioma, anal cancer and colorectal cancer, an estimated 50 to 100 of each tumor type. To collect and store blood samples from patients with gastric cancer, GIST, esophageal cancer, pancreas cancer, hepatocellular cancer, biliary cancer, neuroendocrine, peritoneal mesothelioma, anal cancer and colorectal cancer. To create a database for the collected tissue and allow access to relevant clinical information for current and future protocols. To create tissue microarrays for each gastrointestinal cancer subtype, namely, gastric cancer, GIST, esophageal cancer, pancreas cancer, hepatocellular cancer, biliary cancer, neuroendocrine, peritoneal mesothelioma, anal cancer and colorectal cancer, to facilitate future molecular studies. To grant access to Dr Kindler, Dr. Salgia, and Dr. Catenacci to this database (as it is being acquired) of the coupled patient tissue samples (normal and malignant) and relevant clinical information for the investigation of tyrosine kinases, such as Met and Ron, receptor tyrosine kinase family members, STATs, paxillin, focal adhesion proteins, cell motility/migration proteins, tyrosine/serine/threonine kinase family members, related molecules, and downstream targets implicated in the pathogenesis of GI cancers. Examples of molecular testing include evaluation of DNA mutation, alternative splice variants, protein expression and phosphorylation, and immunohistochemistry on samples. These studies will be correlated with clinical information as stated above.

ELIGIBILITY:
Inclusion Criteria:

* any patient diagnosed with Gastric (stomach) Cancer, Esophageal (foodpipe) Cancer, Pancreas Cancer, Liver Cancer, Biliary (gallbladder) Cancer, Gastrointestinal Stromal Tumor, Peritoneal Mesothelioma (cancer in the lining of the abdomen), Neuroendocrine (of or relating to the cells that release a hormone into the blood in response to a neural stimulus) Tumor, Anal Cancer or Colorectal Cancer cancer that requires you to undergo a surgical or diagnostic procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient having a biopsy or having surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-07-02 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Collect and store blood samples | 1 year
  To collect and store blood samples from patients with gastric cancer, GIST, esophageal cancer, pancreas cancer, hepatocellular cancer, biliary cancer, neuroendocrine, peritoneal mesothelioma, anal cancer and colorectal cancer.
create a database for the collected tissue | 1 year
  To create a database for the collected tissue and allow access to relevant clinical information for current and future protocols.

SECONDARY OUTCOMES:
To create tissue microarrays for each gastrointestinal cancer subtype | 1 year
  To create tissue microarrays for each gastrointestinal cancer subtype, and to facilitate future molecular studies. To grant access to this database (as it is being acquired) of the coupled patient tissue samples (normal and malignant) and relevant clinical information for the investigation of tyrosine kinases, such as Met and Ron, etc., and downstream targets implicated in the pathogenesis of GI cancers. Examples of molecular testing include evaluation of DNA mutation, alternative splice variants, protein expression and phosphorylation, and immunohistochemistry on samples.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Catenacci, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States